#### INFORMED CONSENT FORM – FATHER

Title: Effect of Enhanced Recovery After Cesarean (ERAS) Protocol on Mother-Infant and

Father-Infant Bonding: A Multicenter Randomized Controlled Trial

**Protocol Code:** ERAS-CS-BOND-1

Principal Investigator: Dr. Gökçenur Karakelleoğlu

**Institution:** Istanbul Okan University Hospital

Country: Türkiye

Version: 1.0

Date: November 04, 2025

NCT Number: Not yet Assigned

#### INFORMED CONSENT FORM – FATHER

Study Title: Effect of ERAS Protocol on Father-Infant Bonding

Principal Investigator: Dr. Gökçenur Karakelleoğlu

## 1. Purpose

To evaluate the effect of ERAS on father-infant bonding during the first postpartum week.

#### 2. Procedure

On postpartum day 7, you will complete the PBQ questionnaire (10 minutes). No medical procedure is involved.

#### 3. Risks/Discomfort

No physical risks. Emotional discomfort may occur; you may stop at any time.

#### 4. Benefits

No direct clinical benefit; results may help improve family-centered postpartum care.

## 5. Confidentiality

Data coded, stored for 15 years, no names in publications.

## 6. Voluntary Participation

You may withdraw without any consequences.

# 7. Contact

Dr. Gökçenur Karakelleoğlu

## **Consent Statement**

"I have read this form and voluntarily agree to participate."

Father's Name / Signature / Date

Researcher's Signature / Date